CLINICAL TRIAL: NCT06927154
Title: Comparison of Facet Oscillatory Mobilization and Mobilization With Movement in Chronic Mechanical Neck Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC-01007 Hidayat Ullah
Record Dates: First submitted 2025-04-07; First posted 2025-04-15 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Chronic Mechanical Neck Pain
Keywords: Chronic Mechanical Neck Pain; Facet Oscillatory Mobilization; Mobilization with Movement (MWM)
MeSH Terms: interventions — Movement

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobilization with movement (Experimental)
  Interventions: Other: Mobilization with movement
- Facet joint oscillatory mobilization (Experimental)
  Interventions: Other: Facet joint oscillatory mobilization

INTERVENTIONS:
Other: Mobilization with movement — Group A will receive Mobilization with movement in which therapist manually applies a gentle mobilizing force to the joint while the patient actively performs a movement (2 to 3 sets) 6 to 10 repetitions per set in sitting position. Conventional treatment (TENS (2 to 10 Hz),10 mints, Heating pad, stretching of tight muscles Trapezius and SCM)should be included.
  Other Names: Facet joint oscillatory mobilization Interventions:
  Arms: Mobilization with movement
Other: Facet joint oscillatory mobilization — Group B will receive Facet joint oscillatory mobilization on the cervical spine C2-C7 (6 to 10 repetitions in each session) in the sitting position.Conventional treatment (TENS (2 to 10 Hz) 10 mints, Heating pad, stretching of tight muscles Trapezius and SCM) should be included.
  Other Names: Mobilization with movement
  Arms: Facet joint oscillatory mobilization

SUMMARY:
The study compares Facet Oscillatory Mobilization and Mobilization with Movement in managing chronic mechanical neck pain, aiming to determine the effectiveness of these techniques in pain, range of motion, and disability.

DETAILED DESCRIPTION:
This study will be Conducted as a randomized controlled trial, it will include 32 participants divided into two groups receiving different mobilization techniques along with conventional physical therapy. Outcome measures such as the Numeric Pain Rating Scale (NPRS), Neck Disability Index (NDI), and Inclinometer will be used to assess changes over a two-week intervention period with a follow-up after one month.

ELIGIBILITY:
Inclusion Criteria:

* complaint of Chronic Mechanical neck pain ( more than 6 weeks).
* Neck Disability Index (NDI) score more than 16%
* Age between 35-45 years, Both Male and Female
* NPRS score more than 3-6.
* Recurrent neck pain aggravated at least once in the month.
* Painful Cervical ROM (Flexion less than 80, Extension less than 70, rotation less than 90 to both sides and lateral flexion less than 35 degree.

Exclusion Criteria:

* Cervical radiculopathy
* Cervical canal stenosis
* Severe neurological disorder
* Previous cervical surgery
* Recent history of fall/trauma to the cervical spine.

Ages: 35 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-04-18 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Numeric pain rating scale (NPRS) | Four Weeks
  A subjective pain assessment tool where patients rate their pain intensity on a scale from 0 (no pain) to 10 (worst imaginable pain).
Inclinometer | Four Weeks
  An inclinometer is a device used in physiotherapy to measure joint range of motion (ROM), particularly in the cervical spine. It provides objective and reliable assessments of neck mobility, helping to track progress in patients with chronic mechanical neck pain.
Neck Disability Index (NDI) | Four Weeks
  The NDI is a self-reported questionnaire used to assess the impact of neck pain on daily activities, including personal care, work, sleep, and recreation.

CONTACTS AND LOCATIONS:
Overall Officials: Amnah Anum, MSPT, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Malakand, Chakdara, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: No